## Remotely Supervised Transcranial Direct Current Stimulation for Persistent Posttraumatic Headache

NCT04012853

October 15, 2021

Independent two-tailed t-tests and Fisher Exact tests were used to compare continuous and categorical (respectively) group level demographics, TBI characteristics, and baseline headache features. To investigate measures of safety and tolerability, as well as feasibility and compliance, we compared group differences in self-reported treatment side-effects and intervention attrition using a series of Fisher Exact tests. To assess the efficacy of our RS-tDCS intervention we first investigated within-group changes from baseline using a series of dependent t-tests. Finally, a linear regression model was used to investigate group differences between active and sham RS-tDCS.